CLINICAL TRIAL: NCT02441556
Title: Acute Basilar Artery Occlusion: Endovascular Interventions vs Standard Medical Treatment
Acronym: BEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinfeng Liu (Other)
Responsible Party: Sponsor-Investigator, Xinfeng Liu, Professor and Chairman of Department of Neurology, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JLH-NEURO-2015-001
Record Dates: First submitted 2015-04-16; First posted 2015-05-12 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2016-12

CONDITIONS: Stroke Due to Basilar Artery Occlusion; Acute Cerebrovascular Accidents
Keywords: thrombectomy; rt-PA; stroke; endovascular treatment; randomized
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard medical therapy (Active Comparator): Patients receive standard medical therapy alone.
  Interventions: Other: standard medical therapy
- endovascular + standard medical therapy (Experimental): Patients receive endovascular treatment plus standard medical therapy.
  Interventions: Device: endovascular treatment; Other: standard medical therapy

INTERVENTIONS:
Device: endovascular treatment — The endovascular treatment is comprised of thrombolysis, mechanical thrombectomy, stenting, or a combination of all these approaches. Generally, Solitaire FR is preferred, other devices such as Trevo or future advanced devices can also be considered which will be decided by the executive committee.
  Arms: endovascular + standard medical therapy
Other: standard medical therapy — If the patient meets the criteria for IV rt-PA within 4.5 h of stroke onset, he/she will receive a single alteplase dose of 0.9 mg/kg IV(maximum dose: 90mg), with 10% given as a bolus, followed by continuous IV infusion of the other dose within 1h. All patients will receive standard medical therapy. The standard medical therapy conforms with the current American Heart Association/American Stroke Association guidelines.

SUMMARY:
This trial will provide valuable insights into the safety and efficacy of endovascular treatment for acute ischemic stroke patients with basilar artery occlusion within 8 hours of estimated occlusion time.

DETAILED DESCRIPTION:
This clinical trial is designed to compare the safety and efficacy of endovascular treatment plus standard medical therapy with standard medical therapy alone for acute BA occlusion presented within 8 h of estimated occlusion time. There is only one ongoing clinical trial-Basilar Artery International Cooperation Study (BASICS) (NCT01717755) aimed to evaluate the efficacy and safety of additional intra-arterial treatment after intravenous treatment in 750 patients with BA occlusion, which was anticipated to be completed in Oct 2017. Initiation of intra-arterial therapy should be feasible within 6 hours of estimated time of BA occlusion. And patients are required to have an NIHSS ≥ 10 at time of randomization, and take IV rt-PA, age between 18-85 years old.

In this trial, the investigators did not have age or NIHSS score limit, patients who did not fulfill the requirements for IV rt-PA can also be included into the trial, the investigators also extended the time window to 8 hours which will accelerate the recruitment of potential subjects. In endovascular treatment arm, the time interval between randomization to procedure finish will be controlled within 120 mins. The preparation of endovascular treatment will start immediately after randomization for those eligible patients for IV rt-PA within 4.5 hours after acute stroke onset, with no need to wait for the one-hour rt-PA infusion. A positive trial will suggest substantial clinical benefit from endovascular treatment plus standard medical therapy over standard medical therapy. This trial may provide novel evidence of adopting endovascular treatment for acute patients with BA occlusion, which may consequently advance our current approach for acute stroke treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Acute ischemic stroke consistent with infarction in the basilar artery territory;
3. Basilar artery occlusion confirmed by CTA/MRA/DSA, within 8 hours of estimated occlusion time;
4. Written informed consent from patient or surrogate, if unable to provide consent.

Exclusion Criteria:

1. Computed tomography (CT) or Magnetic Resonance Imaging (MRI) evidence of Cerebral hemorrhage on presentation;
2. Premorbid mRS ≥ 3 points;
3. Currently in pregnant or lactating;
4. Known serious sensitivity to radiographic contrast agents and nitinol metal;
5. Current participation in another investigation drug or device study;
6. Uncontrolled hypertension defined as systolic blood pressure > 185 mmHg or diastolic blood pressure > 110 mmHg that cannot be controlled except with continuous parenteral antihypertensive medication;
7. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency; or oral anticoagulant therapy with INR >1.7 or institutionally equivalent prothrombin time;
8. Baseline lab values: glucose < 50 mg/dl or > 400 mg/dl, platelets <100*109/L, or Hct<25%;
9. Arterial tortuosity that would prevent the device from reaching the target vessel;
10. Life expectancy less than 1 year;
11. History of major hemorrhage in the past 6 months;
12. Angiographic evidence of significant cerebellar mass effect or acute hydrocephalus.
13. Angiographic evidence of bilateral extended brainstem ischemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2015-01; Primary Completion 2017-09-27 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) | at 90 days from randomization
  A score of 0-3 will be considered as the favorable outcome.

SECONDARY OUTCOMES:
mRS score 0-2 | at 90 days from randomization
Change of mRS score(shift analysis) | at 90 days from randomization
Vessel recanalization rate evaluated by CT angiography or MRA | at 24 hours from randomization
PC-ASPECT score on CT/MRI | at 24 hours from randomization
GCS score | at 24 hours from randomization
NIHSS score | at 24 hours from randomization
GCS score | at 5-7 days from randomization
NIHSS score | at 5-7 days from randomization
EuroQol 5D (EQ-5D) | at 90 days from randomization
mortality | at 3 months from randomization
symptomatic intracerebral hemorrhage (ICH) | within 24 hours from randomization
incidence of non-intracerebral hemorrhage complications | at 90 days from randomization
severity of non-intracerebral hemorrhage complications | within 90 days from randomization
incidence of nonbleeding severe adverse events (SAEs) | within 90 days from randomization
severity of nonbleeding severe adverse events (SAEs) | within 90 days from randomization
incidence of procedure and device related complications | within 90 days from randomization
  i.e., vessel perforation, clinically significant groin complications, dissection, arterial occlusion and embolization, etc.
severity of procedure and device related complications | within 90 days from randomization
  i.e., vessel perforation, clinically significant groin complications, dissection, arterial occlusion and embolization, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Xinfeng Liu, Doctor, Study Chair — Departmnet of Neurology, Jinling Hospital
Locations (44):
- China (44):
  - 123rd Hospital of The People's Liberation Army, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - the First Affiliated Hospital of An'hui Medical University, Hefei, Anhui
  - the First People's Hospital of Huainan, Huainan, Anhui
  - Lu'an Affiliated Hospital of Anhui Medical University, Lu'an, Anhui
  - Yijishan Hospital of Wannan Medical College, Wuhu, Anhui
  - Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Fuzhou General Hospital of Nanjing Military Region, Fuzhou, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - 175th hospital of PLA, the Affiliated Southeast Hospital of Xiamen University, Xiamen, Fujian
  - Affiliated Zhongshan Hospital of Xiamen University, Xiamen, Fujian
  - Guangdong No.2 Provincial People's Hospital, Guangzhou, Guangdong
  - The Chinese Armed Police Force Guangdong Armed Police Corps hospital, Guangzhou, Guangdong
  - Maoming People's Hospital, Maoming, Guangdong
  - Shenzhen Nanshan Hospital, Shenzhen, Guangdong
  - Henan Provincial People's Hospital,Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Zhongshan Hospital, Wuhan, Hubei
  - Wuhan No.1 Hospital, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - Jinling Hospital, Medical School of Nanjing University, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - 101st hospital of PLA, Wuxi, Jiangsu
  - the Second Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - the Third People's Hospital of Yancheng, Yancheng, Jiangsu
  - Yangzhou No.1 People's Hospital, Yangzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - the First People's Hospital of Yangzhou， Yangzhou University, Yangzhou, Jiangsu
  - Yangzhou Hongquan Hospital, Yangzhou, Jiangsu
  - Linyi People's Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Taian City Central Hospital, Taian, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Chengdu Military General Hospital, Chengdu, Sichuan
  - Sichuan People's Hospital, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - the First People's Hospital of Hangzhou,Nanjing Medical University, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Lishui Central Hospital, Lishui, Zhejiang
  - Xinqiao Hospital, the Third Military Medical University, Chongqing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schonewille WJ, Wijman CA, Michel P, Rueckert CM, Weimar C, Mattle HP, Engelter ST, Tanne D, Muir KW, Molina CA, Thijs V, Audebert H, Pfefferkorn T, Szabo K, Lindsberg PJ, de Freitas G, Kappelle LJ, Algra A; BASICS study group. Treatment and outcomes of acute basilar artery occlusion in the Basilar Artery International Cooperation Study (BASICS): a prospective registry study. Lancet Neurol. 2009 Aug;8(8):724-30. doi: 10.1016/S1474-4422(09)70173-5. Epub 2009 Jul 3. PMID 19577962
- [Background] National Institute of Neurological Disorders and Stroke rt-PA Stroke Study Group. Tissue plasminogen activator for acute ischemic stroke. N Engl J Med. 1995 Dec 14;333(24):1581-7. doi: 10.1056/NEJM199512143332401. PMID 7477192
- [Background] Hacke W, Kaste M, Bluhmki E, Brozman M, Davalos A, Guidetti D, Larrue V, Lees KR, Medeghri Z, Machnig T, Schneider D, von Kummer R, Wahlgren N, Toni D; ECASS Investigators. Thrombolysis with alteplase 3 to 4.5 hours after acute ischemic stroke. N Engl J Med. 2008 Sep 25;359(13):1317-29. doi: 10.1056/NEJMoa0804656. PMID 18815396
- [Background] Saqqur M, Uchino K, Demchuk AM, Molina CA, Garami Z, Calleja S, Akhtar N, Orouk FO, Salam A, Shuaib A, Alexandrov AV; CLOTBUST Investigators. Site of arterial occlusion identified by transcranial Doppler predicts the response to intravenous thrombolysis for stroke. Stroke. 2007 Mar;38(3):948-54. doi: 10.1161/01.STR.0000257304.21967.ba. Epub 2007 Feb 8. PMID 17290031
- [Background] Ciccone A, Valvassori L, Nichelatti M, Sgoifo A, Ponzio M, Sterzi R, Boccardi E; SYNTHESIS Expansion Investigators. Endovascular treatment for acute ischemic stroke. N Engl J Med. 2013 Mar 7;368(10):904-13. doi: 10.1056/NEJMoa1213701. Epub 2013 Feb 6. PMID 23387822
- [Background] Broderick JP, Palesch YY, Demchuk AM, Yeatts SD, Khatri P, Hill MD, Jauch EC, Jovin TG, Yan B, Silver FL, von Kummer R, Molina CA, Demaerschalk BM, Budzik R, Clark WM, Zaidat OO, Malisch TW, Goyal M, Schonewille WJ, Mazighi M, Engelter ST, Anderson C, Spilker J, Carrozzella J, Ryckborst KJ, Janis LS, Martin RH, Foster LD, Tomsick TA; Interventional Management of Stroke (IMS) III Investigators. Endovascular therapy after intravenous t-PA versus t-PA alone for stroke. N Engl J Med. 2013 Mar 7;368(10):893-903. doi: 10.1056/NEJMoa1214300. Epub 2013 Feb 7. PMID 23390923
- [Background] Kidwell CS, Jahan R, Gornbein J, Alger JR, Nenov V, Ajani Z, Feng L, Meyer BC, Olson S, Schwamm LH, Yoo AJ, Marshall RS, Meyers PM, Yavagal DR, Wintermark M, Guzy J, Starkman S, Saver JL; MR RESCUE Investigators. A trial of imaging selection and endovascular treatment for ischemic stroke. N Engl J Med. 2013 Mar 7;368(10):914-23. doi: 10.1056/NEJMoa1212793. Epub 2013 Feb 8. PMID 23394476
- [Background] Smith WS, Sung G, Saver J, Budzik R, Duckwiler G, Liebeskind DS, Lutsep HL, Rymer MM, Higashida RT, Starkman S, Gobin YP; Multi MERCI Investigators; Frei D, Grobelny T, Hellinger F, Huddle D, Kidwell C, Koroshetz W, Marks M, Nesbit G, Silverman IE. Mechanical thrombectomy for acute ischemic stroke: final results of the Multi MERCI trial. Stroke. 2008 Apr;39(4):1205-12. doi: 10.1161/STROKEAHA.107.497115. Epub 2008 Feb 28. PMID 18309168
- [Background] Nogueira RG, Lutsep HL, Gupta R, Jovin TG, Albers GW, Walker GA, Liebeskind DS, Smith WS; TREVO 2 Trialists. Trevo versus Merci retrievers for thrombectomy revascularisation of large vessel occlusions in acute ischaemic stroke (TREVO 2): a randomised trial. Lancet. 2012 Oct 6;380(9849):1231-40. doi: 10.1016/S0140-6736(12)61299-9. Epub 2012 Aug 26. PMID 22932714
- [Background] Saver JL, Jahan R, Levy EI, Jovin TG, Baxter B, Nogueira RG, Clark W, Budzik R, Zaidat OO; SWIFT Trialists. Solitaire flow restoration device versus the Merci Retriever in patients with acute ischaemic stroke (SWIFT): a randomised, parallel-group, non-inferiority trial. Lancet. 2012 Oct 6;380(9849):1241-9. doi: 10.1016/S0140-6736(12)61384-1. Epub 2012 Aug 26. PMID 22932715
- [Background] Berkhemer OA, Fransen PS, Beumer D, van den Berg LA, Lingsma HF, Yoo AJ, Schonewille WJ, Vos JA, Nederkoorn PJ, Wermer MJ, van Walderveen MA, Staals J, Hofmeijer J, van Oostayen JA, Lycklama a Nijeholt GJ, Boiten J, Brouwer PA, Emmer BJ, de Bruijn SF, van Dijk LC, Kappelle LJ, Lo RH, van Dijk EJ, de Vries J, de Kort PL, van Rooij WJ, van den Berg JS, van Hasselt BA, Aerden LA, Dallinga RJ, Visser MC, Bot JC, Vroomen PC, Eshghi O, Schreuder TH, Heijboer RJ, Keizer K, Tielbeek AV, den Hertog HM, Gerrits DG, van den Berg-Vos RM, Karas GB, Steyerberg EW, Flach HZ, Marquering HA, Sprengers ME, Jenniskens SF, Beenen LF, van den Berg R, Koudstaal PJ, van Zwam WH, Roos YB, van der Lugt A, van Oostenbrugge RJ, Majoie CB, Dippel DW; MR CLEAN Investigators. A randomized trial of intraarterial treatment for acute ischemic stroke. N Engl J Med. 2015 Jan 1;372(1):11-20. doi: 10.1056/NEJMoa1411587. Epub 2014 Dec 17. PMID 25517348
- [Background] Mattle HP, Arnold M, Lindsberg PJ, Schonewille WJ, Schroth G. Basilar artery occlusion. Lancet Neurol. 2011 Nov;10(11):1002-14. doi: 10.1016/S1474-4422(11)70229-0. PMID 22014435
- [Background] Jauch EC, Saver JL, Adams HP Jr, Bruno A, Connors JJ, Demaerschalk BM, Khatri P, McMullan PW Jr, Qureshi AI, Rosenfield K, Scott PA, Summers DR, Wang DZ, Wintermark M, Yonas H; American Heart Association Stroke Council; Council on Cardiovascular Nursing; Council on Peripheral Vascular Disease; Council on Clinical Cardiology. Guidelines for the early management of patients with acute ischemic stroke: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Mar;44(3):870-947. doi: 10.1161/STR.0b013e318284056a. Epub 2013 Jan 31. PMID 23370205
- [Derived] Liu X, Dai Q, Ye R, Zi W, Liu Y, Wang H, Zhu W, Ma M, Yin Q, Li M, Fan X, Sun W, Han Y, Lv Q, Liu R, Yang D, Shi Z, Zheng D, Deng X, Wan Y, Wang Z, Geng Y, Chen X, Zhou Z, Liao G, Jin P, Liu Y, Liu X, Zhang M, Zhou F, Shi H, Zhang Y, Guo F, Yin C, Niu G, Zhang M, Cai X, Zhu Q, Chen Z, Liang Y, Li B, Lin M, Wang W, Xu H, Fu X, Liu W, Tian X, Gong Z, Shi H, Wang C, Lv P, Tao Z, Zhu L, Yang S, Hu W, Jiang P, Liebeskind DS, Pereira VM, Leung T, Yan B, Davis S, Xu G, Nogueira RG; BEST Trial Investigators. Endovascular treatment versus standard medical treatment for vertebrobasilar artery occlusion (BEST): an open-label, randomised controlled trial. Lancet Neurol. 2020 Feb;19(2):115-122. doi: 10.1016/S1474-4422(19)30395-3. Epub 2019 Dec 9. PMID 31831388
- [Derived] Liu X, Xu G, Liu Y, Zhu W, Ma M, Xiong Y, Zi W, Dai Q, Leung T, Yan B, Davis S, Liebeskind DS, Pereira VM, Nogueira RG; BEST Trial Investigators. Acute basilar artery occlusion: Endovascular Interventions versus Standard Medical Treatment (BEST) Trial-Design and protocol for a randomized, controlled, multicenter study. Int J Stroke. 2017 Oct;12(7):779-785. doi: 10.1177/1747493017701153. Epub 2017 Mar 31. PMID 28361616